CLINICAL TRIAL: NCT01378949
Title: Psoas Compartment Block Versus Fascia Iliaca Block After Total Hip Arthroplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: A. Stav, Hillel Yaffe Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2259-11-HYMC
Record Dates: First submitted 2011-06-19; First posted 2011-06-23 (Estimated); Last update posted 2011-06-23 (Estimated); Status verified 2011-06

CONDITIONS: Pain
Keywords: pain score
MeSH Terms: conditions — Pain | interventions — Bupivacaine; Morphine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- PsCB Group (Active Comparator): Ultrasound-Guided Psoas Compartment Block will be used in patients for pain relief after THA
  Interventions: Drug: Bupivacaine
- FICB Group (Active Comparator): Ultrasound-Guided Fascia Iliaca Compartment Block will be used in patients for pain relief after THA
  Interventions: Drug: Bupivacaine
- Patient-Controlled Analgesia (Active Comparator): Patient-controlled analgesia will be used for pain relief after THA
  Interventions: Drug: Morphine

INTERVENTIONS:
Drug: Bupivacaine — Bupivacaine 0.5% with adrenaline 5 mcg/cc
  Arms: FICB Group; PsCB Group
Drug: Morphine — Morphine 1 mg/cc
  Arms: Patient-Controlled Analgesia

SUMMARY:
A psoas compartment block has been used with good results for postoperative pain relief after total hip arthroplasty (THA). However, case reports describing serious complications after the use of this block, have been reported. The fascia iliaca compartment block (FICB) has been shown to be a reliable block for postoperative pain relief for procedures and injuries involving the hip. The investigators have not found any literature that has compared these two blocks. This study will compare the two blocks when used for post-operative pain relief after THA.

ELIGIBILITY:
Inclusion Criteria:

* ASA Class I-III
* Patients undergoing THA for osteoarthritis

Exclusion Criteria:

* Skin infections adjacent to block site
* Allergy to local analgesics
* Patient unable to understand visual analogue scale (VAS)

Ages: 45 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2011-09; Primary Completion 2013-09 (Estimated); Study Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
Pain score of patients who have been given FICB for post-operative pain relief after THA | 3 days

CONTACTS AND LOCATIONS:
Locations (1):
- Hillel Yaffe Medical Center, Hadera, Israel